CLINICAL TRIAL: NCT01021696
Title: The Impact of Pain on Behavioural Disturbances in Patients With Moderate and Severe Dementia. A Cluster Randomized Trial
Brief Title: Pain in Patients With Dementia and Behavioural Disturbances
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Bergen (Other)
Collaborators: The Research Council of Norway (Other)
Responsible Party: Bettina Sandgathe Husebo, Department of Public Health and Primary Health Care, University of Bergen
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2008-007490-20
Record Dates: First submitted 2009-11-27; First posted 2009-11-30 (Estimated); Last update posted 2011-08-10 (Estimated); Status verified 2010-11

CONDITIONS: Dementia; Pain; Agitation
Keywords: Dementia; Nursing home; Pain treatment; Pain assessment; Agitation
MeSH Terms: conditions — Dementia; Pain; Psychomotor Agitation; Agnosia | interventions — Acetaminophen; Morphine; Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Treatment as usual (No Intervention): Control group
- Paracetamol (Active Comparator): Intervention group
  Interventions: Drug: Paracetamol
- Morphine (Active Comparator): Intervention group, individual pain treatment
  Interventions: Drug: Morphine
- Buprenorphine plaster (Active Comparator): Intervention group, individual pain treatment
  Interventions: Drug: Buprenorphine plaster
- Pregabalin (Active Comparator): Intervention group, individual pain treatment
  Interventions: Drug: Pregabalin

INTERVENTIONS:
Drug: Paracetamol — Paracetamol Max. dose: 3g/d
  Other Names: Individual pain treatment
  Arms: Paracetamol
Drug: Morphine — Morphine ret. Tab. 5mgx2/d; max. dose:10mgx2/d
  Other Names: Individual pain treatment
  Arms: Morphine
Drug: Buprenorphine plaster — 5ųg/h, change each 7.day; max. dose: 10ųg/h
  Other Names: Individual pain treatment
  Arms: Buprenorphine plaster
Drug: Pregabalin — 25mgx1/d; max 300mg/d
  Other Names: individual pain treatment
  Arms: Pregabalin

SUMMARY:
In nursing homes (NHs) 80% of the patients have dementia, between 60%-80% exhibit behavioural disturbances (BPSD), and more than 60% have pain. Both pain and BPSD is more common in those with severe dementia. Since older persons with dementia have less communicative skills, suffer from more pain and exhibit more agitation, pain may be a contributing factor in these patients. More than 40% of patients with BPSD are treated with neuroleptics despite described side-effects. There is an urgent need to investigate the impact of individual pain management on BPSD in patients with dementia.

It was hypothesized that

* pain increase BPSD in patients with dementia
* individual pain treatment decrease BPSD in patients with dementia

DETAILED DESCRIPTION:
We intend to conduct an eight weeks, multi-centre, rater-blinded, cluster randomized, and parallel-group trial, with follow up after four weeks. We will choose cluster randomizing by practical reasons. 920 NH patients were screened and 352 patients with moderate or severe dementia and BPSD were included. The treatment period is 8 weeks, with further follow after four weeks.

The primary outcome measure will be reduction in aggression and agitation as well as other items which are measured by means of CMAI (Cohen Mansfield Agitation Inventory). Secondary outcome are reduction in NPI-NH-subscale agitation/aggression and other items which are measured by the Neuropsychiatric Inventory, Nursing Home Version (NPI-NH). Further, we want to evaluate the concomitant use of acute medication. Additionally, Activities of Daily Living function (ADL) and MIni Mental State Examination (MMSE) will be used as secondary outcome measure.

Pain in patients with dementia will be assessed and followed by the MOBID-2 Pain Scale (secondary outcome measure). MOBID-2 Pain Scale is a staff-administered behavioural instrument for assessment pain in older persons with dementia with god validity and reliability (Husebo 2008, 2009). MOBID-2 is based on patient's pain behaviour in connection with standardised, guided movements of different body part, and pain behaviour related to internal organs, head and skin. Additionally, pain will be registered by pain diagnoses, -etiology, and -duration. The MOBID-2 score is derived from caregiver in a clinical bedside situation during morning care.

Adverse events will be recorded and evaluated throughout the study as the primary assessment of safety and tolerability.

Inclusion criteria: Patients of either gender, 60 years of age or older, living in a nursing home (NH) diagnosed moderate or severe dementia measured by the Functional Assessment Staging (FAST) and MMSE, and BPSD in form of agitation / aggression as measured by subscale of NPI-NH and CMAI.

Exclusion criteria: Patients without cognitive impairment and without BPSD. Patients with hepatic or renal failure or diseases that make it impossible to follow the study schedule.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 and older
* Residing in the NHs for at least 4 weeks
* Dementia according to Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) (American Psychiatric Association 1994), FAST score > 4 (Hughes 1982).
* Clinically relevant BPSD, operationally defined as CMAI score ≥ 39 or higher or/and at least one week history of agitation or aggression (Koss 1997).
* Written, informed consent provided by the participant (if they have capacity) or assent (if they do not have capacity) and a written proxy informed consent from a legally authorized representative empowered to make health-related decisions for the potential study participant.

Exclusion Criteria:

* Clinician responsible for care, or study clinician considers that the patient suffers from any physical condition, which would make participation in the trial distressing or likely to increase suffering
* Advanced severe medical disease/disorder with expected survival less than 6 months or that could interfere with participation
* Psychosis or other severe mental disorder prior to dementia diagnosis;
* Severe aggression (≥8) on item 3 of the NPI subscale, with aggression as the predominant symptom
* Schizophrenia, schizoaffective disorder and bipolar disorder
* Uncontrolled epilepsy
* Severe liver impairment
* Renal failure, as measured by or equivalent to an estimated creatinine clearance of < 50mL/min/1.73m,
* Severe injury or anaemia (Hb < 8.5 mmol/l), comatose state, current enrolment in another experimental protocol.
* Known allergy or adverse reaction to Paracetamol, Morphine ret, Buprenorphine plaster or pregabalin

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 352 (Actual)
Dates: Start 2009-11; Primary Completion 2010-07 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Cohen-Mansfield Agitation Inventory - long form (CMAI) | CMAI will be used during the screening/inclusion process, at week 2, 4, 8, and 12.
  CMAI has 29-item (max. score 203) to assess agitated behaviours in NH-patients. A six-point rating scale assesses the frequency with which patients manifest BPSD evaluating 29 agitated behaviours, ranging from never, less than once a week, but still occurring, once or twice a week, several times a week, once or twice a day, several times a day or several times an hour. Items are presented in four factors: I Aggressive behaviour; II Physical non-aggressive behaviour; III Verbally agitated behavior, IV hiding and hoarding. Ratings are based on face-to-face interviews with caregivers.

SECONDARY OUTCOMES:
Neuropsychiatric Inventory - Nursing Home Version (NPI-NH) | NPI will be used during the inclusion process, at week 2, 4, 8, and 12.
  NPI is a caregiver based interview (10 min.), assessing 10 BPSD and 2 neurovegetative areas with total score and subscales for: delusion, hallucination, agitation, depression, anxiety, disinhibition apathy, irritability, aberrant motor activity, sleep, appetite. Frequency, severity, and caregiver's distress are measured. The NH-version will be used, recently validated in Norwegian (AGS Panel 1998). A higher score reflects increased frequency and severity of the disturbances.
Activity of Daily Living function (ADL) | ADL assessment will be used during clinical investigation related to the inclusion prosess and at week 8
  ADL assess physical function. Rating includes activities like feeding, moving, personal toilet, and dressing higher values indicating higher levels of activities of daily functioning and independency (Sheikh 1979). The scale includes 10 items (0-20 score). The ADL score is derived from caregiver interview. Administration of the ADL takes approximately 5 minutes.
Mini Mental State Examination | Screening/clinical investigation and week 8
  The MMSE is a 30-point mental status examination scale that enables cut-off differentiation for levels of severity of cognitive impairment (Folstein 1975). Cut point for moderate dementia: <20. The question consist of several orientation question (10 points), registration and recall task (6), attention task (5), three stage command (3), two naming task (2), repetition task (1), reading comprehension task (1), written sentence (1), and a visual construction (1). The test takes 15 minutes to administer and the patient is asked the questions directly by the examiner.
Mobilisation-Observation-Behavior-Intensity-Dementia-2 (MOBID-2) Pain Scale | Screening/clinical investigation, week 2,4,8,12
  MOBID-2 Pain Scale is a staff-administered behavioural instrument for assessment pain in older persons with dementia (Husebo 2008a). MOBID-2 is based on patient's pain behaviour in connection with standardised, guided movements of different body part, and pain behaviour related to internal organs, head and skin. Additionally, pain will be registered by pain diagnoses, -etiology, and -duration. The MOBID-2 score is derived from caregiver in a clinical bedside situation during morning care. Administration of the MOBID-2 takes approximately 5 minutes.
Functional Assessment Staging (FAST) | Screening and week 8
  FAST describes a continuum of seven stages and sub stages from normality to most severe dementia (Hughes 1982). Moderate to severe dementia is consistent with Fast stage of 5 or 6 or 7. Stage 5 is defined as moderately severe cognitive decline, with deficient performance in activities of daily living such as choosing proper clothing and maintaining hygiene. Stage 6 is defined as severe cognitive decline with incontinence and decreased ability to clothe, bathe, toilet oneself, severely limited speech, vocabulary, emotional expression. FAST score is derived from caregiver interview (5 min).
Adverse events (AE) and serious adverse event (SAE) | week 2,4,8
  Safety and tolerability assessments will consist of monitoring and recording all adverse events (AE) and serious adverse events (SAE) and the regular monitoring of vital signs (BP, puls); AE and SAE registration and report is related to each patient, each medication each centre with reportation to the Norwegian Medicines Agency (study code EUDRACTNR. 2008-007490-20).

CONTACTS AND LOCATIONS:
Overall Officials: Rolv Terje Lie, PhD, Study Director — University of Bergen, Norway; Bettina S. Husebo, MD, PhD, Study Chair — University of Bergen, Norway; Dag Aarsland, MD, Phd, Principal Investigator — University of Bergen, Norway; Clive Ballard, MD, PhD, Principal Investigator — King's College London
Locations (18):
- Norway (18):
  - Knarvik Nursing Home, Knarvik, Horadland
  - Aastveit Nursing Home, Åstveit, Hordaland
  - Dormkirkehjemmet, Bergen, Hordaland
  - Fantoft Omsorgssenter, Bergen, Hordaland
  - Bergen Red Cross Nursing Home, Bergen, Hordaland
  - Solsletten Sykehjem, Bergen, Hordaland
  - Mildeheimen, Bergen, Hordaland
  - Søreide Nursing Home, Bergen, Hordaland
  - Lindas bu- og servicecentre, Isdalstø, Hordaland
  - Saata bu og servicecentre, Isdalstø, Hordaland
  - Lyngbøtunet Nursing Home, Laksevåg, Hordaland
  - Odinsvei Nursing Home, Nesttun, Hordaland
  - Ovsttunheimen, Nesttun, Hordaland
  - Slaathaug Nursing Home, Hafrsfjord, Rogaland
  - Rovik Nursing Home, Sandnes, Rogaland
  - Sola Nursing Home, Sola, Rogaland
  - Blidensol Nursing Home, Stavanger, Rogaland
  - Tasta Nursing Home, Stavanger, Rogaland

REFERENCES:
- [Background] Husebo BS. [Pain assessment in dementia]. Tidsskr Nor Laegeforen. 2009 Oct 8;129(19):1996-8. doi: 10.4045/tidsskr.08.0660. Norwegian. PMID 19823204
- [Background] Husebo BS, Strand LI, Moe-Nilssen R, Husebo SB, Ljunggren AE. Pain behaviour and pain intensity in older persons with severe dementia: reliability of the MOBID Pain Scale by video uptake. Scand J Caring Sci. 2009 Mar;23(1):180-9. doi: 10.1111/j.1471-6712.2008.00606.x. Epub 2009 Jan 20. PMID 19192240
- [Background] Husebo BS, Strand LI, Moe-Nilssen R, Borgehusebo S, Aarsland D, Ljunggren AE. Who suffers most? Dementia and pain in nursing home patients: a cross-sectional study. J Am Med Dir Assoc. 2008 Jul;9(6):427-33. doi: 10.1016/j.jamda.2008.03.001. Epub 2008 Jun 2. PMID 18585645
- [Background] Husebo BS, Strand LI, Moe-Nilssen R, Husebo SB, Snow AL, Ljunggren AE. Mobilization-Observation-Behavior-Intensity-Dementia Pain Scale (MOBID): development and validation of a nurse-administered pain assessment tool for use in dementia. J Pain Symptom Manage. 2007 Jul;34(1):67-80. doi: 10.1016/j.jpainsymman.2006.10.016. Epub 2007 May 23. PMID 17509814
- [Derived] Griffioen C, Husebo BS, Flo E, Caljouw MAA, Achterberg WP. Opioid Prescription Use in Nursing Home Residents with Advanced Dementia. Pain Med. 2019 Jan 1;20(1):50-57. doi: 10.1093/pm/pnx268. PMID 29136228
- [Derived] Aasmul I, Husebo BS, Flo E. Staff Distress Improves by Treating Pain in Nursing Home Patients With Dementia: Results From a Cluster-Randomized Controlled Trial. J Pain Symptom Manage. 2016 Dec;52(6):795-805. doi: 10.1016/j.jpainsymman.2016.07.004. Epub 2016 Aug 12. PMID 27524403
- [Derived] Habiger TF, Flo E, Achterberg WP, Husebo BS. The Interactive Relationship between Pain, Psychosis, and Agitation in People with Dementia: Results from a Cluster-Randomised Clinical Trial. Behav Neurol. 2016;2016:7036415. doi: 10.1155/2016/7036415. Epub 2016 May 9. PMID 27247487
- [Derived] Husebo BS, Ballard C, Fritze F, Sandvik RK, Aarsland D. Efficacy of pain treatment on mood syndrome in patients with dementia: a randomized clinical trial. Int J Geriatr Psychiatry. 2014 Aug;29(8):828-36. doi: 10.1002/gps.4063. Epub 2013 Dec 19. PMID 24806873
- [Derived] Husebo BS, Ballard C, Cohen-Mansfield J, Seifert R, Aarsland D. The response of agitated behavior to pain management in persons with dementia. Am J Geriatr Psychiatry. 2014 Jul;22(7):708-17. doi: 10.1016/j.jagp.2012.12.006. Epub 2013 Apr 20. PMID 23611363
- [Derived] Husebo BS, Ballard C, Sandvik R, Nilsen OB, Aarsland D. Efficacy of treating pain to reduce behavioural disturbances in residents of nursing homes with dementia: cluster randomised clinical trial. BMJ. 2011 Jul 15;343:d4065. doi: 10.1136/bmj.d4065. PMID 21765198